CLINICAL TRIAL: NCT05733494
Title: Cross-Cultural Adaptation and Validation of the Italian Version of the Clinical Assessment of Dysphagia in Neurodegeneration (CADN)
Brief Title: Cross Cultural Validation of the Italian Version of the Clinical Assessment of Dysphagia in Neurodegeneration
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Micol Castellari, Speech-Language Pathologist, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: CE2622
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Swallowing Disorder; Dysphagia; Neuro-Degenerative Disease
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with neurodegenerative disease: Patients with neurodegenerative disease
  Interventions: Other: Administration of Clinical Assessment of Dysphagia in Neurodegeneration (CADN)

INTERVENTIONS:
Other: Administration of Clinical Assessment of Dysphagia in Neurodegeneration (CADN) — the CADN will be administrated to each patient at the enrolment

SUMMARY:
The English version of the "Clinical Assessment of Dysphagia in Neurodegeneration" (CADN), represents a rapid and valid clinical assessment tool for dysphagia in neurodegenerative population.

Currently, there is no validated tool in Italian specific for the clinical assessment of dysphagia in neurodegenerative disease with strong psychometric characteristics.

The present study aims to translate and validate the Italian version of CADN in neurodegenerative population. Psychometric properties will be measured.

DETAILED DESCRIPTION:
Most of patients with a neurodegenerative disease will develop swallowing impairments (dysphagia) during their disease progression (up to 80%- 100% in Parkinson disease and Amyotrophic Lateral Sclerosis).

Dysphagia is associated with serious clinical complications, particularly regarding loss of life quality, insufficient medication intake, malnutrition, dehydration, and aspiration with subsequent pneumonia, which is the leading cause of death in this population.

Early detection and measurement of dysphagia trough validated and standardized procedures plays a fundamental role in the clinical practice. Clinical assessment by a speech language pathologist (SLP) can provide early identification of dysphagia and its severity and direct clinical decision making.

The English version of the "Clinical Assessment of Dysphagia in Neurodegeneration" (CADN), represents a rapid and valid clinical assessment tool for dysphagia in neurodegenerative population.

Currently, there is no validated tool in Italian specific for the clinical assessment of dysphagia in neurodegenerative disease with strong psychometric characteristics.

The present study aims to translate and validate the Italian version of CADN in neurodegenerative population.

The study will be carried out in two phases:

1. Forward and back translation
2. Validation process

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of neurodegenerative disease according to the respective consensus criteria
* >18 years old
* able to provide informed consent
* able to follow simple instructions
* capable of sitting upright for anamnesis and examination for at least 20 min (in chair or wheelchair)

Exclusion Criteria:

* history of stroke
* surgery to the head or neck
* radiotherapy in the last 12 months
* dysphagia resulting from other known causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with neurodegenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment of Dysphagia in Neurodegeneration (CADN) | at the enrolment
  Clinical assessment tool administrated by a Speech Language Pathologist. The CADN is composed by a clinical case history and a consumption part for a total of 11 item. Severity scores for each item range from 0 (no impairment) to 4 (severe impairment).
Clinical Assessment of Dysphagia in Neurodegeneration (CADN) | at 24 hours from enrolment
  Clinical assessment tool administrated by a Speech Language Pathologist. The CADN is composed by a clinical case history and a consumption part for a total of 11 item. Severity scores for each item range from 0 (no impairment) to 4 (severe impairment).

SECONDARY OUTCOMES:
Fiberoptic Endoscopic Evaluation of Swallowing (FEES) | At the enrolment
  Instrumental examination, gold standard for the assessment of dysphagia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Milano, Italy